CLINICAL TRIAL: NCT06147141
Title: Effectiveness and Mechanism of Online Peer Companion Intervention on Children With Autism Spectrum Disorders: A Randomized Controlled Trial
Brief Title: Effectiveness and Mechanism of Online Peer Companion Intervention on Children With Autism Spectrum Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, YinyinZang, School of Psychological and Cognitive Sciences, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPCI on Children with ASD
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Peer-Mediated Intervention; Children
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Online Peer Companion Intervention group (OPCI) and Wait-List Group (WLG)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Peer Companion Intervention group (OPCI) (Experimental): experimental group
  Interventions: Behavioral: Online Peer Companion Intervention
- Wait-List Group (WLG) (Placebo Comparator): control group
  Interventions: Behavioral: Wait-List

INTERVENTIONS:
Behavioral: Online Peer Companion Intervention — Ordinary children would be paired with ASD children before the interventions. Dyads in the OPCI would have a total of 12 sessions within two months, each lasting 30-60 minutes. The longest interval between two sessions couldn't exceed two weeks. Researchers would recommend a series of companion themes for children to choose from (e.g., daily sharing and drawing). Ordinary children and ASD children need to discuss activities that are of mutual interest before each session. A researcher assistant would be online to ensure the normal development of the interventions and be responsible for video recording of the exchanges at the beginning of each session. Except for extreme circumstances, he or she would turn off the video and sound throughout the process and withdraw soon. During the interventions, parents would play a supporting role when children express needs without over-involvement.
  Arms: Online Peer Companion Intervention group (OPCI)
Behavioral: Wait-List — Dyads in the WLG would only participate in preliminary training and measurement during the implementation of the intervention. After completing the post-test, this study will implement the same online peer companionship intervention.
  Arms: Wait-List Group (WLG)

SUMMARY:
The goal of this interventional study was to examine the effectiveness and mechanism of online peer companion intervention (OPCI) on the social abilities and mental health of ASD children. The main questions it aims to answer are:

1. Whether OPCI is effective on the social abilities and mental health of ASD children;
2. What impact does OPCI have on the social abilities and mental health of ordinary children;
3. What impact does OPCI have on the mental health of both children's parents;
4. What are the mechanisms of OPCI on ASD children.

ELIGIBILITY:
Inclusion Criteria of ASD Children:

* 7-15 years old and diagnosed as mild ASD;
* Basic ability to speak independently and fluently communicate with peers;
* Could use mobile phones, tablets, computers, or other electronic devices for this online intervention.

Exclusion Criteria of ASD Children:

* Diagnosed as moderate or severe ASD;
* Unable or unwilling to communicate with peers independently
* No phones or other alternative electronic devices for the intervention Inclusion

Criteria of Ordinary Children:

* 9-18 years old with normal development, no diagnosis of ASD, learning disabilities, ADHD, and other mental disorders;
* Lively and outgoing, able to assume the role of topic organizer in communication with peers;
* Could use mobile phones, tablets, computers, or other electronic devices for this online intervention.

Exclusion Criteria of Ordinary Children

* Diagnosis of ASD or other neurodevelopmental and mental disorders;
* Introverted or unwilling to play with peer ASD children
* No phones or other alternative electronic devices for the intervention

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Social Behavior of ASD Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention
  We examined the effectiveness of OPCI on the social behavior of ASD participants through parent-report Social Responsiveness Scale (SRS).
Mental Health of ASD Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention
  We examined the effectiveness of OPCI on the mental health of ASD participants through the parent-report 25-item Revised Child Anxiety and Depression Scale (RCADS)

SECONDARY OUTCOMES:
Mental Health of Ordinary Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention) or only measure at pre-test, post-test and follow-up
  We examined the effectiveness of OPCI on the mental health of ordinary children participants through some self-report and parent-report scales, including the 25-item Revised Child Anxiety and Depression Scale (RCADS), Connor-Davidson resilience scale (CD-RISC), and so on.
Social Ability of Ordinary Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention
  We explored the effectiveness of OPCI on the social ability of ordinary children participants through self-report and parent-report Social Skills Rating Systems (SSRS)
Mental Health of Parents | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention) or only measure at pre-test, post-test and follow-up.
  We examined the effectiveness of OPCI on the mental health of both children's parents through some self-report scales, including the General Anxiety Disorder Scale-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), Connor-Davidson resilience scale (CD-RISC), and so on.

OTHER OUTCOMES:
Intervention Process Screen Recording Coding | each session
  We coded the screen recording of interventions to explore the effectiveness and influencing factors of OPCI. Videos for each dyad will be conducted by a trained undergraduate student. This work will be carried out under the guidance and supervision of a professional clinical psychologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No